CLINICAL TRIAL: NCT06554015
Title: Prospective Longitudinal Study of Heylo™ for People Living With a Stoma
Status: Recruiting | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP370
Record Dates: First submitted 2024-07-02; First posted 2024-08-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to longitudinally evaluate the usage and long-term benefits of the CE-marked device, Heylo™, a digital leakage notification system for people with intestinal stomas. The system, which includes a smartphone application, an adhesive sensor layer, and a Bluetooth transmitter, notifies users of changes in their baseplate status, potentially reducing stoma effluent leakage and improving quality of life. The physical Heylo™ device, is part of the Coloplast Charter telehealth service.

ELIGIBILITY:
Inclusion Criteria:

1. Are you at least 18 years old? [Yes/No]
2. Do you have an ileostomy or a colostomy? [Yes/No]
3. Have you used Heylo™ for less than seven days? [Yes/No]

Exclusion Criteria:

1) Do you have a stoma reversal planned (surgery date within the next 6 months)? Yes/No]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outside this investigation, stoma patients eligible for the Heylo™ device prescription, will be onboarded to Heylo™ by stoma care nurses.
  Subjects for this study will be identified through their Heylo™ app activation. A minimum of 100 subjects will be enrolled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | one year
  Stoma-related QoL measured by the Emotional Leakage Impact score (domain 1 of OLI) at baseline (0 months), 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

REFERENCES:
- [Derived] Vestergaard M, Gunning A, Mather R, Hansen HD, Ajslev TA. Impact of a Digital Leakage Notification System on Leakage, Quality of Life, Healthcare Resource Utilisation, and Work Productivity: Interim Results from a Longitudinal Real-World Study in the UK. J Clin Med. 2026 Jan 14;15(2):663. doi: 10.3390/jcm15020663. PMID 41598602